CLINICAL TRIAL: NCT00830466
Title: A Randomized Trial to Study Combined Pulsed Dye Laser and Rapamycin Treatment of Port Wine Stain Birthmarks.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J S Nelson, M.D., Ph.D.,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20086383
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Port Wine Stain
Keywords: port wine stain
MeSH Terms: conditions — Port-Wine Stain | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser and rapamycin versus laser alone (Experimental): Laser and rapamycin versus laser alone
  Interventions: Drug: Laser and rapamycin versus laser alone

INTERVENTIONS:
Drug: Laser and rapamycin versus laser alone — Laser and rapamycin versus laser alone

SUMMARY:
The researchers want to collect data on safety and efficacy of combined pulsed dye laser and rapamycin to improve fading/blanching of port wine stain birthmarks as compared to pulsed dye laser alone, which is the current standard of care.

This single center pilot and feasibility study will have a target enrollment of 40 port wine stain subjects at the Beckman Laser Institute and Medical Clinic, University of California, Irvine.

DETAILED DESCRIPTION:
The study will offer two different approaches to the treatment of port wine stain birthmarks.

Study Group Number 1: Port wine stain treated by the pulsed dye laser alone, which is the current standard of care: 20 subjects.

Study Group Number 2: Port wine stain treated by combined pulsed dye laser and rapamycin: 20 subjects.

The researchers want to collect data on safety and efficacy of combined pulsed dye laser and rapamycin to improve fading/blanching of port wine stain birthmarks as compared to pulsed dye laser alone, which is the current standard of care. Twenty subjects will have their entire port wine stain birthmark treated by pulsed dye laser alone. Twenty subjects will have their entire port wine stain birthmark treated by combined pulsed dye laser and rapamycin, which is a drug that prevents the formation of blood vessels in the skin. Safety will be evaluated by searching for any local effects such as injury to the skin or systemic effects such as abnormal blood and/or urine studies. Efficacy will be determined by objectively measuring and comparing the port wine stain fading/blanching responses for the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Port wine stain suitable for comparison testing.
* Age > 13 years of age or older; minor will be accompanied in the room by parents or guardians during laser treatment.
* Apparent good health as documented by medical history.
* Ability to understand and carry out subject instructions.
* Women of childbearing potential must have a negative urinary pregnancy test prior to being started on rapamycin.
* Women of child bearing potential must agree to use a medically acceptable method of contraception throughout the study and for 3 months following discontinuation of rapamycin.

Exclusion Criteria:

* Inability to understand and carry out instructions.
* Pregnancy.
* Abnormal blood or urine tests
* History of cancer.
* History of high cholesterol, lipids or liver disease.
* Allergy to macrolide drugs (e.g., erythromycin).
* Any therapy within the previous two months to the proposed port wine stain treatment sites.
* Current participation in any other investigational drug evaluation.
* Concurrent use of known photosensitizing drugs.
* Concurrent use of immunosuppressive drugs or steroids.
* Concurrent use of any of the following medications: antifungals, antiepileptics, protease inhibitors, cimetidine, cisapride, clarithromycin, dannzol, diltiazem, erythromycin, metoclopramide, rifabutin, rifampin, rifapetine, troleandomycin, or verapamil.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Improved port wine stain fading/blanching after laser treatment | 24 weeks
  Efficacy will be determined by objectively measuring and comparing the port wine stain fading/blanching responses for subjects treated with combined pulsed dye laser and rapamycin versus pulsed dye laser alone

CONTACTS AND LOCATIONS:
Overall Officials: J. Stuart Nelson, M.D.,Ph.D., Principal Investigator — Beckman Laser Institute and Medical Clinic, University of California Irvine
Locations (1):
- Beckman Laser Institute and Medical Clinic, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Undecided